CLINICAL TRIAL: NCT04167527
Title: Endovascular Therapy for Low NIHSS Ischemic Strokes
Acronym: ENDOLOW
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of Calgary (Other); University of Cincinnati (Other); Heidelberg University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Raul Gomes Nogueira, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00107210
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Ischemia
Keywords: Immediate Mechanical Thrombectomy; Initial medical management; Large vessel occlusion; Efficacy; Safety
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate mechanical thrombectomy(iMT) (Experimental): Treatment initiation within 8 hours of symptom onset. Arterial puncture and revascularization will be performed using EmboTrap II Retriever. The procedure will be completed within two hours of arterial access.
  Interventions: Device: Immediate mechanical thrombectomy(iMT) using EmboTrap Revascularization Device
- Initial medical management (iMM) (Active Comparator): Standard medical therapy based on current AHA (American Heart Association) guidelines. Rescue mechanical thrombectomy (rMT) is allowed for patients initially assigned to iMM if they suffer major neurological worsening that clearly requires an intra-arterial intervention in the judgment of the treating team.
  Interventions: Combination Product: Initial medical management (iMM)

INTERVENTIONS:
Device: Immediate mechanical thrombectomy(iMT) using EmboTrap Revascularization Device — Treatment initiation is defined as the date and time of arterial puncture. Femoral artery puncture will occur within 45 minutes of randomization and no longer than 90 minutes after the completion of the qualifying imaging. It must occur before 8 hours since the subject was last known well.The initial procedure will be performed using only the EmboTrap II Retriever for the first two passes, and a third pass is encouraged. Date and time of arterial puncture, revascularization, and procedure end will be recorded. It is expected that the interventional procedure will be completed within two hours of arterial access.
  All subjects, regardless of randomization arm, will receive best medical management based on current American Heart Association, Canadian, or European guidelines according to their geographic location.
  Other Names: EmboTrap III
  Arms: Immediate mechanical thrombectomy(iMT)
Combination Product: Initial medical management (iMM) — Patients will receive standard medical therapy based on current AHA guidelines. For patients who are treated with intravenous tissue plasminogen activator (rtPA), the sites' post-rtPA protocol will be followed. Rescue mechanical thrombectomy (rMT) is allowed for patients initially assigned to iMM if they suffer major neurological worsening that clearly requires an intra-arterial intervention in the judgment of the treating team.
  All subjects, regardless of randomization arm, will receive best medical management based on current American Heart Association, Canadian, or European guidelines according to their geographic location.
  Arms: Initial medical management (iMM)

SUMMARY:
This study will test the hypothesis that patients presenting within 8 hours of onset with cerebral ischemia in the setting of proximal large vessel occlusions (LVO) and low baseline NIHSS scores (0-5) will have better 90-day clinical outcomes (mRS distribution) with immediate mechanical thrombectomy (iMT) compared to initial medical management (iMM).

DETAILED DESCRIPTION:
Currently, the vast majority of these patients do not receive immediate vessel imaging with either CT- or MR-angiography. However, acute ischemic stroke patients with low NIHSS who harbor a large vessel occlusion (LVO) later decline in 20-40% of cases, and/or have underappreciated impairments related to their relatively mild strokes. Similarly, LVO patients presenting with a transient ischemic attack (TIA) are under increased risk of clinical deterioration. Such patients with apparent good collateral circulation, and hence a substantial perfusion of the vascular territory of the occluded large artery, likely have the most to gain from endovascular revascularization. At the same time, this collateral perfusion may allow for more frequent recanalization, either spontaneously or by intravenous (IV) rtPA. Experience with immediate mechanical thrombectomy (iMT) in the LVO mild stroke target population is limited.

This study will test the hypothesis that patients presenting within 8 hours of onset with cerebral ischemia in the setting of proximal large vessel occlusions (LVO) and low baseline NIHSS scores (0-5) will have better 90-day clinical outcomes (mRS distribution) with immediate mechanical thrombectomy (iMT) compared to initial medical management (iMM).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Acute ischemic stroke based on clinical diagnosis (NIHSS 0-5) and presence of an objective neurological deficit
3. Patients eligible for intravenous rt-PA should receive this therapy as soon as possible and no later than 4.5 hours from symptom onset
4. Proximal Intracranial Artery Occlusion on Imaging by NCCT/CTA or MRI/MRA showing complete occlusion of the intracranial ICA, M1, or an "M1-like" M2 vessel with or without tandem cervical lesion. Notably, "M1-like" M2 vessel occlusions are defined functionally for the trial as following:

   1. On CTA: Occlusion of both branches after MCA division (both M2s occluded) or occlusion of the larger diameter M2 branch . In case of trifurcations, either the two largest M2 branches are occluded or the occluded M2 has a larger diameter than the combined diameter of the two other M2s . Notably, the M2 origins are defined by the first branching point in the MCA other than the anterior temporal artery rather than by anatomic landmarks (e.g., horizontal versus insular location).

      or
   2. If mCTA or CTP performed (optional): a M2 occlusion which supplies a large proportion of the MCA territory by evidence of either:

   i. The bulk (>2/3) of the MCA territory has evidence of delayed washout on multiphase CT or ii. Perfusion imaging shows a hypoperfusion lesion volume involving a significant proportion of the MCA territory defined as Tmax >4 sec lesion of ≥100 mL
5. Baseline Infarct Core of either:

   1. Baseline ASPECTS ≥6 on non-contrast CT (NCCT), or
   2. Baseline Infarct Core Volume of < 70cc on either CTP (Volume of rCBF <30%) or DWI if quantitative software tools are available (neither test is mandatory for study)

Exclusion Criteria:

1. NIHSS ≥6
2. Any sign of intracranial hemorrhage on baseline CT/MR (SDH/SAH/ICH)
3. Any imaging findings suggestive of futile recanalization in the judgment of the local investigator
4. High degree of suspicion of intracranial arterial disease (ICAD), such as evidence of multifocal ICAD
5. Premorbid disability (mRS ≥3)
6. Inability to randomize within 8 hours of last known well
7. Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS
8. Baseline blood glucose of <50 mg/dL (2.78 mmol) or >400 mg/dL (22.20 mmol)
9. Known coagulation disorders as defined as platelet count <100,000/uL
10. Known renal failure as defined as serum creatinine levels > 3.0 mg/dL
11. Presumed septic embolus or suspicion of bacterial endocarditis
12. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.
13. Participation in another investigational treatment study in the previous 30 days
14. Intubation and mechanical ventilation prior to study enrollment is medically indicated
15. History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
16. Site investigator does not have equipoise towards the ideal treatment concept (thrombectomy vs. best medical management)
17. Known pregnancy
18. Prisoner or incarceration
19. Known acute symptomatic COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
90-day Global Disability Assessed Via the Blinded Evaluation of Modified Rankin Score (Ordinal Shift Analysis). | 90-day
  The distribution of the modified Rankin Scale (mRS) is assessed by structured assessment. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
Symptomatic intracranial hemorrhage (sICH) within 36 hours comparing the two treatment arms | 36 hours
  Symptomatic intracranial hemorrhage (sICH) within 36 hours post treatment imaging scan, using SITS-MOST criteria, consisting of the presence of parenchymal hematoma type 2 (PH2) on neuroimaging associated with 4-point decline in NIHSS from baseline to 24 hours
Symptomatic intracerebral hemorrhage within 96 hours comparing the two treatment arms | 96 hours
  Symptomatic intracerebral hemorrhage is defined as local or remote parenchymal hemorrhage type 2, subarachnoid hemorrhage, and/or intraventricular hemorrhage within 96 hours post-randomization, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 hour, or leading to death

SECONDARY OUTCOMES:
Shift in distribution of the 90-day mRS with levels 5-6 combined (0;1;2;3;4;5-6) comparing the two treatment arms | 90-day
  The distribution of the 90-day modified Rankin Scale (mRS) with levels 5-6 combined (0;1;2;3;4;5-6) is assessed by structured assessment. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
Number of patients with good outcome comparing the two treatment arms | 90-day
  Good outcome is defined by a score of 0-2 on the 90-day mRS. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
Number of patients with excellent outcome comparing the two treatment arms arms | 90-day
  Excellent outcome is defined by a score 0-1 on the 90-day mRS. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire.
Number of patients with early Neurologic Deterioration (END) comparing the two treatment arms | 24 hours post randomization
  Early Neurologic Deterioration (END) is defined as an increase in NIHSS of ≥4 points. NIH Stroke Scale/Score (NIHSS) is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items.
Health-related quality of life EQ-5D score comparing the two treatment arms | 90-day
  EQ-5D is a standardized instrument measuring health-related quality of life. The EQ-5D consists of a descriptive system and the EQ VAS.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number.
Infarct volume | 24 hours post randomization
  Infarct volume is a direct measurement of one of the final pathologic steps leading to the clinical deficits caused by an ischemic stroke.Final infarct volume derived from MR imaging.
Self-reported mental and physical health PROMIS Global-10 score | 90-day
  Mental and physical health will be assessed using PROMIS Global-10. The PROMIS Global-10 short form consists of 10 items that assess general domains of health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.Scores are converted to a T-Score metric.
Self-reported PROMIS Fatigue score | 90-day
  The PROMIS Fatigue assesses a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities.
  Each question has five response options ranging in value from one to five.To find the total raw score, values of the response to each question will be summed up. Total raw score will be transformed into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Number of patients with intracranial hemorrhages using the Heidelberg Bleeding definition comparing the two treatment arms | 90-day
  Intracranial hemorrhages will be defined using the Heidelberg Bleeding criteria.
Mortality rate within 90 days comparing the two treatment arms | 90-day
  Mortality rate will be calculated.
Instrumental Activities of Daily Living (IADL) | 90-day
  Instrumental Activities of Daily Living (IADLs) are activities related to independent living. The IADL scale covers eight functional domains: using the telephone, shopping, food preparation, housekeeping, laundry, transport, medication, and finances. Participants are scored according to their highest level of functioning in categories, and summary score ranges from 0 (low function, dependent) to 8 (high function, independent).

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — Emory University
Locations (34):
- United States (26):
  - Providence Little Company of Mary Medical Center, Torrance, California
  - Baptist Health Jacksonville FL, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Grady Health System (non-CRN), Atlanta, Georgia
  - Rush University Medical Center: University Neurosurgery, Chicago, Illinois
  - Advocate Aurora Health, Downers Grove, Illinois
  - Indiana University, Bloomington, Indiana
  - University of Iowa, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Health Care Corporation, Grand Blanc, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - JFK Neurosciences Center, Edison, New Jersey
  - Thomas Jefferson University, Woodbury, New Jersey
  - Albany Medical Center, Albany, New York
  - University at Buffalo Neurosurgery/ Kaleida Health, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State Wexner Medical Center, Columbus, Ohio
  - Riverside Medical Center, OhioHealth Research Institute, Columbus, Ohio
  - Prisma Health-Upstate, Greenville, South Carolina
  - Semmes Murphey Foundation, Memphis, Tennessee
  - Texas Tech University Health Sciences Center at El Paso, El Paso, Texas
  - VHS-Harlingen Hospital Company dba Valley Baptist Medical Center-Harlingen, Harlingen, Texas
- Canada (6):
  - University of Calgary and Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Germany (2):
  - Universitäts Klinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Ludwig Maximilian University, Department of Neurology, München, Bavaria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article will be available after de-identification and in accordance with applicable laws and regulations. Other limited data sets may be provided as governed by ENDOLOW Publications SOP and in accordance with ICMJE.
Supporting Information: Study Protocol
Time Frame: Data will become available beginning 1 year after publication of the primary analysis.
Access Criteria: After primary analysis publication, site investigators will have the opportunity to contribute to secondary, tertiary and quaternary analysis of the data and publication. Additionally, after 1 year, non-investigator researchers may submit requests to the publications committee for additional analysis after providing a methodologically sound proposal. Proposals can be sent to ENDOLOW-CCC@emory.edu. Data Transfer Agreements may apply.

REFERENCES:
- [Derived] Seners P, Cereda CW. Thrombectomy in Stroke With a Large Vessel Occlusion and Mild Symptoms: "Striving to Better, Oft We Mar What's Well?". Stroke. 2023 Sep;54(9):2276-2278. doi: 10.1161/STROKEAHA.123.044205. Epub 2023 Aug 1. No abstract available. PMID 37526012
- [Derived] Feil K, Matusevicius M, Herzberg M, Tiedt S, Kupper C, Wischmann J, Schonecker S, Mengel A, Sartor-Pfeiffer J, Berger K, Dimitriadis K, Liebig T, Dieterich M, Mazya M, Ahmed N, Kellert L. Minor stroke in large vessel occlusion: A matched analysis of patients from the German Stroke Registry-Endovascular Treatment (GSR-ET) and patients from the Safe Implementation of Treatments in Stroke-International Stroke Thrombolysis Register (SITS-ISTR). Eur J Neurol. 2022 Jun;29(6):1619-1629. doi: 10.1111/ene.15272. Epub 2022 Feb 19. PMID 35122371